CLINICAL TRIAL: NCT07118332
Title: Psilocybin as a Treatment for Chronic Pain in Smokers
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry • MEDPSY Psych Divisions- SATU, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Psilocybin
Record Dates: First submitted 2025-07-23; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Smokers With Chronic Pain
Keywords: cigarettes; pain
MeSH Terms: conditions — Pain | interventions — Psilocybin; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin 25mg (Experimental)
  Interventions: Drug: Psilocybin (drug)

INTERVENTIONS:
Drug: Psilocybin (drug) — 25mg of Psilocybin will be given to all subject

SUMMARY:
The purpose of this study is to understand whether psilocybin therapy is safe and well tolerated in improving chronic pain and increasing motivation to quit smoking for people who have chronic pain and smoke cigarettes. Psilocybin is a psychedelic drug and the active ingredient in "magic mushrooms." Psilocybin is currently being studied in clinical trials but has no current medical use in the United States. Some studies have shown that a dose of psilocybin can help people quit smoking. Other studies have shown that a dose of psilocybin may improve certain chronic pain conditions, such as migraine headaches. We believe that it may also be helpful for people who smoke and have chronic pain, but this has not been tested yet.

DETAILED DESCRIPTION:
This will be an open-label pilot study examining the feasibility and potential efficacy of psilocybin in individuals who smoke and have chronic pain. Following the screening visit, the potential participants will have 1) an adaptation/preparation session, 2) a treatment session, and 3) two post-treatment follow-up sessions: 1 and 4 weeks after the treatment session. During study participation, participants will also complete surveys 4 times per day on a mobile device for 5 weeks (1 week before the treatment session and 4 weeks post-treatment session).

General Procedures: Potential participants will undergo extensive medical and psychiatric screening to minimize the risk of study participation. Psilocybin will be administered as a 25 mg oral dose under close medical and psychiatric monitoring.

For the 24 hours before the treatment session, subjects will be asked to abstain from consuming alcoholic beverages and any illicit drugs, verified by urine drug screening and breathalyzer. Non-compliant subjects will be rescheduled or discharged from the study if they are repeatedly non-compliant. Subjects will be instructed to drink their typical number of caffeinated beverages and smoke cigarettes as usual to minimize caffeine and tobacco withdrawal, which could confound the study measures. Subjects will be instructed not to eat for 4 hours before the treatment sessions because a light snack will be provided before the beginning of the session, and lunch will be provided at the end.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 21 to 65 years, who have been smoking tobacco cigarettes daily cigarettes for at least a year (confirmed with urine cotinine strips indicating smoking status (28)
* not seeking treatment at the time of the study for tobacco use.
* endorsement of bothersome or high-impact chronic non-cancer pain per the Graded Pain Scale - Revised (29);
* in good health as verified by medical history, screening examination, and screening laboratory tests; and
* body mass index (BMI) between 18 to 35 because there is limited information on the safety of psilocybin in individuals outside this range.
* for women, not pregnant as determined by pregnancy screening, nor breastfeeding, and using acceptable birth control methods (e.g., oral contraceptives).

Exclusion Criteria:

* History of major medical disorders (e.g., diabetes, epilepsy, kidney or liver diseases, heart rhythm problems, heart failure, hypertension with BP greater than 140/90mmHg, history of cerebrovascular problems, severe asthma, etc.).
* lifetime history of schizophrenia, bipolar disorder, dissociative disorders, or borderline personality disorder, current major depressive episode, or PTSD.
* first- or second-degree relatives with a history of bipolar disorder or schizophrenia.
* suicide attempt or ideation in the past year.
* regular use of certain psychotropic medications (antidepressants, antipsychotics, mood stabilizers or anxiolytics) that are deemed to have the potential for adverse effects or drug reactions with psilocybin including SSRIs and MAO inhibitors.
* current untreated moderate or severe substance use disorder for any other recreational or prescription drugs other than nicotine.
* known sensitivity or intolerability to psilocybin.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
SAFTEE scale | Day 1 and Day 7
  The SAFTEE will be administered before and after each session to monitor adverse events from the study medications. The SAFTEE has been used in many pharmacotherapy trials (52) and includes possible side effects of study medications.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided